CLINICAL TRIAL: NCT05743413
Title: Evaluation of the Effect of Rehabilitation Using the Armeo Spring Device on Improving the Quality of Motion of Upper Extremity in Patients in the Sub-acute Stage After Stroke and Its Correlation With the Rate of Improvement in the Quality of Life After Completing Rehabilitation
Brief Title: Improving the Quality of Life of Stroke Patients Using the Armeo Spring Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital Ostrava (Other)
Collaborators: University of Ostrava (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FNO-KRTL-01
Record Dates: First submitted 2023-02-14; First posted 2023-02-24 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Ischemic Stroke
Keywords: ischemic stroke; rehabilitation; Armeo Spring therapy; quality of life
MeSH Terms: conditions — Ischemic Stroke

STUDY DESIGN:
Intervention Model Description: The study participants will be enrolled into two parallel groups.
Masking Description: No masking will be used in the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Armeo Spring (Experimental): Study subjects randomized into this group will undergo physiotherapy sessions using the Armeo Spring device.
  Interventions: Procedure: Armeo Spring physiotherapy
- Standard physiotherapy (Active Comparator): Study subjects randomized into this control group will undergo standard physiotherapy sessions.
  Interventions: Procedure: Standard physiotherapy

INTERVENTIONS:
Procedure: Armeo Spring physiotherapy — Study subjects will undergo physiotherapy sessions using the Armeo Spring device.
  Arms: Armeo Spring
Procedure: Standard physiotherapy — Study subjects will undergo standard physiotherapy sessions.
  Arms: Standard physiotherapy

SUMMARY:
The main goal will be to evaluate the effect of improving the quality of movement of the upper limb (using an evaluation exercise in the software of the Armeo Spring device) on the development of the quality of life after stroke using a standardized generic and specific questionnaire.

The secondary outcome will be to evaluate changes in self-sufficiency using a test of daily activities modified by the Frenchay test of daily activities.

DETAILED DESCRIPTION:
The research follows on from a pilot study that took place at the Department of Rehabilitation and Sports Medicine, University Hospital Ostrava from 4/2022 to 9/2022. It has a prospective monocentric randomized trial design. Patients will be randomized into parallel groups - intervention and control groups.

A prospective monocentric randomized study lasting 8 months at the Department of Rehabilitation and Sports Medicine, University Hospital Ostrava. The study design is parallel with a test and control arm. Patients will be divided into an intervention (tested) group A with therapy on Armeo Spring and a control group B with conventional therapy, using a random number generator, where odd numbers represent arm A and even numbers represent arm B. A randomization table randomly allocates patients to therapy according to their order of entry into the study.

ELIGIBILITY:
Inclusion Criteria:

* history of stroke
* age over 18 years
* Modified Rankin Scale (mRS) of 2-3
* moderate paresis of the upper extremity (individuals with shoulder/elbow muscle test values in the range of 3-1)
* cardiovascular stability

Exclusion Criteria:

* age under 18 years
* severe cognitive or sensory deficit and non-cooperation
* severe osteoporosis
* impaired skin integrity in the trunk and upper limbs
* cardiovascular instability
* unstable fractures
* acute inflammatory diseases

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2023-08-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Change of upper extremity function - A GOAL | 3 weeks
  Exercise A Goal is an assessment exercise that aims to evaluate the accuracy of the patient's gross motor movements. After placing the pointer on the base, the target will appear. The patient must try to catch the target in a perfectly linear motion and then stay exactly in the center of the target for 3 seconds.
Change of upper extremity function - HPR | 3 weeks
  The HPR value (hand path ratio) is used to evaluate the quality of the patient's movement. It is calculated by dividing the length of the path of the patient's hand by the distance between the points to be grasped in the exercises. A perfectly straight movement has an HPR value of 1. An HPR value of 2 means that the path length of the patient's hand was twice as long as the shortest line connecting the points.
Change of upper extremity function - deviation | 3 weeks
  The deviation shows the distance of the pointer to the center point of the target s, so it is the accuracy value on the target. The value describes the patient's ability to meet positional accuracy. A perfect match between the indicator and the resulting target position represents a deviation value of 0. A deviation value of 2 means that the patient missed the target position by 2 cm.
Change of upper extremity function - variability | 3 weeks
  Variability represents the standard deviation of the points on the track from their average coordinates and is therefore a value of accuracy on target. The value describes the patient's ability to maintain a steady position. Maintaining a perfectly stable position has a variability value of 0. A variability of 2 cm means that 68% of the points on the track are within 2 cm.
Quality of Life - EQ-5D | 3 weeks
  These are standardized questionnaires, i.e. providing exact results of measuring the quality of life in various domains of health status. The EQ-5D group of questionnaires is used worldwide and is one of the most widely used scales in healthcare. It has been certified and translated into many languages. Its use is validated by recent meta-analyses. The questionnaires monitor a total of 5 domains of quality of life - mobility, self-care, normal activities, pain, discomfort, anxiety and depression.

SECONDARY OUTCOMES:
Modified Frenchay Scale (MFS) test | 3 weeks
  The Modified Frenchay Scale (MFS) measures active upper limb function in hemiparesis based on a video review of 10 everyday living tasks, each rated on a 10-point visual analogic scale. Six tasks are bimanual and four are unimanual performed with the paretic hand.
The Barthel Index (BI) | 3 weeks
  The Barthel Index (BI) measures the extent to which somebody can function independently and has mobility in their activities of daily living (ADL) i.e. feeding, bathing, grooming, dressing, bowel control, bladder control, toileting, chair transfer, ambulation and stair climbing.

CONTACTS AND LOCATIONS:
Overall Officials: Šárka Anežka Čechová, MD, Principal Investigator — University Hospital Ostrava
Locations (1):
- University Hospital Ostrava, Ostrava, Moravian-Silesian Region, Czechia

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data available to other researchers. The data may be provided upon request.